CLINICAL TRIAL: NCT02284685
Title: A Novel Intervention Promoting Eating Disorder Treatment Among College Students
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sarah Ketchen Lipson, PhD Candidate, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: F037058; 1F31MH105149-01 (NIH)
Record Dates: First submitted 2014-11-03; First posted 2014-11-06 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Eating Disorders
Keywords: Mental Health Services
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- A (opt-out, loss, social norming) (Experimental): Students in this intervention arm must opt-out of receiving linkage to eating disorder resources on their campus; messages include social norming (statistics comparing their rates of eating disorder symptoms to national averages on widely-used and clinically validated screening tools); and messages frame the negative consequences (losses) of not seeking-help for current disordered eating symptoms. The intervention ('A Novel Intervention Promoting Eating Disorder Treatment among College Students') is this version of the email messages (opt-out, loss, social norming).
  Interventions: Behavioral: Promoting Eating Disorder Treatment among College Students
- B (opt-out, gain, social norming) (Experimental): Students in this intervention arm must opt-out of receiving linkage to eating disorder resources on their campus; messages include social norming (statistics comparing their rates of eating disorder symptoms to national averages on widely-used and clinically validated screening tools); and messages frame the benefits of seeking-help for current disordered eating symptoms. The intervention ('A Novel Intervention Promoting Eating Disorder Treatment among College Students') is this version of the email messages (opt-out, gain, social norming).
  Interventions: Behavioral: Promoting Eating Disorder Treatment among College Students
- C (opt-out, loss, no social norming) (Experimental): Students in this intervention arm must opt-out of receiving linkage to eating disorder resources on their campus; messages do not include social norming (statistics comparing their rates of eating disorder symptoms to national averages on widely-used and clinically validated screening tools); and messages frame the negative consequences (losses) of not seeking-help for current disordered eating symptoms. The intervention ('A Novel Intervention Promoting Eating Disorder Treatment among College Students') is this version of the email messages (opt-out, loss, no social norming).
  Interventions: Behavioral: Promoting Eating Disorder Treatment among College Students
- D (opt-out, gain, no social norming) (Experimental): Students in this intervention arm must opt-out of receiving linkage to eating disorder resources on their campus; messages do not include social norming (statistics comparing their rates of eating disorder symptoms to national averages on widely-used and clinically validated screening tools); and messages frame the benefits of seeking-help for current disordered eating symptoms. The intervention ('A Novel Intervention Promoting Eating Disorder Treatment among College Students') is this version of the email messages (opt-out, gain, no social norming).
  Interventions: Behavioral: Promoting Eating Disorder Treatment among College Students
- E (opt-in, loss, social norming) (Experimental): Students in this intervention arm must opt-in to receiving linkage to eating disorder resources on their campus; messages include social norming (statistics comparing their rates of eating disorder symptoms to national averages on widely-used and clinically validated screening tools); and messages frame the negative consequences (losses) of not seeking-help for current disordered eating symptoms. The intervention ('A Novel Intervention Promoting Eating Disorder Treatment among College Students') is this version of the email messages (opt-in, loss, social norming).
  Interventions: Behavioral: Promoting Eating Disorder Treatment among College Students
- F (opt-in, gain, social norming) (Experimental): Students in this intervention arm must opt-in to receiving linkage to eating disorder resources on their campus; messages include social norming (statistics comparing their rates of eating disorder symptoms to national averages on widely-used and clinically validated screening tools); and messages frame the benefits of seeking-help for current disordered eating symptoms. The intervention ('A Novel Intervention Promoting Eating Disorder Treatment among College Students') is this version of the email messages (opt-in, gain, social norming).
  Interventions: Behavioral: Promoting Eating Disorder Treatment among College Students
- G (opt-in, loss, no social norming) (Experimental): Students in this intervention arm must opt-in to receiving linkage to eating disorder resources on their campus; messages do not include social norming (statistics comparing their rates of eating disorder symptoms to national averages on widely-used and clinically validated screening tools); and messages frame the negative consequences (losses) of not seeking-help for current disordered eating symptoms. The intervention ('A Novel Intervention Promoting Eating Disorder Treatment among College Students') is this version of the email messages (opt-in, loss, no social norming).
  Interventions: Behavioral: Promoting Eating Disorder Treatment among College Students
- H (opt-in, gain, no social norming) (Experimental): Students in this intervention arm must opt-in to receiving linkage to eating disorder resources on their campus; messages do not include social norming (statistics comparing their rates of eating disorder symptoms to national averages on widely-used and clinically validated screening tools); and messages frame the benefits of seeking-help for current disordered eating symptoms. The intervention ('A Novel Intervention Promoting Eating Disorder Treatment among College Students') is this version of the email messages (opt-in, gain, no social norming).
  Interventions: Behavioral: Promoting Eating Disorder Treatment among College Students

INTERVENTIONS:
Behavioral: Promoting Eating Disorder Treatment among College Students — Online intervention designed to identify and increase help-seeking among undergraduates with previously undiagnosed/untreated eating disorders

SUMMARY:
Eating disorders (EDs) have the highest rate of mortality of any mental illness. On U.S. college campuses, an estimated 80% students with clinically significant ED symptoms do not receive treatment. There are likely more than one million students whose EDs go untreated in any given year. Left untreated EDs typically become more severe and refractory to treatment. Given the impact of EDs on mental and physical health and the connection therein with social, academic, and economic outcomes, an effective intervention to increase rates of treatment utilization would have broad societal effects extending well beyond the campus setting. This study is an online intervention designed to identify and increase help-seeking among undergraduates with previously undiagnosed/untreated EDs.

DETAILED DESCRIPTION:
Eating disorders (EDs) have the highest rate of mortality of any mental illness. ED age of onset coincides with the undergraduate years (ages 18-25). As such, colleges provide access to a large, epidemiologically vulnerable population and present a unique opportunity for intervention. On college campuses, 14% of female and 4% of male students screen positive for clinically significant EDs. An estimated 80% of these students do not receive treatment. Left untreated EDs typically become more severe and refractory to treatment. Help-seeking interventions typically focus on minimizing stigma, improving knowledge, and addressing other barriers emphasized by classic theories of health behavior. On the whole, these interventions have failed to increase treatment utilization for the vast majority of students with ED symptoms. Innovative approaches are urgently needed to narrow the ED treatment gap on college campuses.

The proposed study builds on the most comprehensive research to date on mental health service utilization in college populations, which the Principal Investigator of this study (PI) has developed with her faculty advisor. Findings reveal new insight into the ED treatment gap: students with untreated EDs report not seeking help for reasons such as lack of time, lack of perceived need, ambivalence about the severity of need, belief that the problem will resolve itself without treatment, and a desire to deal with issues "on my own." These reasons imply a lack of urgency but not necessarily a strong resistance to receiving treatment. In similar health contexts (e.g., for diet/exercise, use of preventative care), behavioral economic interventions have produced positive results by addressing several cognitive biases, including the default bias (individuals 'go with the flow' of preset options) and the sign effect (losses (negative outcomes) are substantially more psychologically costly than gains (positive outcomes)). The present intervention study addresses these biases in an effort to increase service use among undergraduate students with untreated ED symptoms (as identified in an online screen).

In a 12-week study, the study team is using a factorial design to test the effects of three intervention components: peer norming, default option, and sign effect. The intervention components are delivered via email messaging. To address the default bias, email messages reframe treatment use as an opt-out (as opposed to opt-in) behavior, thus nudging students to seek help. Students are able to check a box to opt out of receiving treatment linkage. Those who do not opt-out receive, without any purposeful action, continued assistance connecting to treatment. For the sign effect, messages emphasize the negative consequences of untreated EDs to engender urgency. Students in conditions with peer norming see how their levels of eating disorder symptoms (results from widely-used, validated measures included in the baseline survey) compare with average symptom levels among other undergraduates (with data taken from national surveys previously conducted by the study team). Follow-up data is being collected at weeks 6 and 12. Intervention components are operationalized in electronic messages delivered over 12-weeks (anticipated: January-May 2015).

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate at participating university
* Untreated symptoms of an eating disorder (as identified in an online screen)

Exclusion Criteria:

* Less than 18 years of age
* Studying abroad during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1149 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Help-seeking behavior (Use of services (e.g., counseling/therapy) for eating and body image issues) | 12 weeks
  Use of services (e.g., counseling/therapy) for eating and body image issues

SECONDARY OUTCOMES:
Predictors of help-seeking behavior (e.g., perceived need/urgency, knowledge, attitudes, intentions to seek help) | 12 weeks
  Predictors of help-seeking behavior (e.g., perceived need/urgency, knowledge, attitudes, intentions to seek help)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K Lipson, MEd, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - University of Michigan, Ann Arbor, Michigan
  - Bard College, Annandale-on-Hudson, New York
  - Appalachian State University, Boone, North Carolina
  - Mercyhurst University, Erie, Pennsylvania